CLINICAL TRIAL: NCT02786576
Title: Effectiveness of Adalimumab in Moderate to Severe HidrAdenitis SuppuRativa Patients - a Multi cOuNtry studY in Real Life Setting - HARMONY Study
Brief Title: Effectiveness of Adalimumab in Moderate to Severe HidrAdenitis SuppuRativa Patients - a Multi cOuNtry studY in Real Life Setting
Acronym: HARMONY
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-769
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2019-09

CONDITIONS: Hidradenitis Suppurativa
Keywords: Moderate to Severe Hidradenitis Suppurativa; Adalimumab
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving adalimumab: Hidradenitis Suppurativa (HS) participants receiving adalimumab

SUMMARY:
This study will assess the effects of adalimumab treatment in moderate to severe Hidradenitis Suppurativa (HS) patients in the real world setting. The objectives of this study are to estimate the effectiveness of adalimumab treatment on disease severity, to estimate the impact of adalimumab treatment on patients' quality of life, psychological effect, work productivity and healthcare resource utilization and to describe treatment practices over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe Hidradenitis Suppurativa
* The decision to treat with adalimumab (Humira) is made by the physician in accordance with the local label (Summary of Product Characteristics; product label) prior to any decision to approach the participant to participate in this study
* Participants willing to be involved in the study and to sign patient authorization form to use and disclose personal health information (or informed consent, where applicable)

Exclusion Criteria:

* Participants in a clinical interventional study
* Participants treated with adalimumab prior to baseline visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hidradenitis Suppurativa (HS) participants receiving adalimumab
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with moderate to severe Hidradenitis Suppurativa (HS) who achieve a clinical response | At Week 12
  Clinical response is evaluated by using the Hidradenitis Suppurativa clinical response measure (HiSCR)

SECONDARY OUTCOMES:
Proportion of participants with moderate to severe HS who achieve a clinical response | Up to week 52
  Clinical response is evaluated by using the Hidradenitis Suppurativa clinical response measure (HiSCR)
Changes from baseline in Dermatology Quality of Life Index (DLQI) | From Week 0 to Week 52
  Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (83):
- Austria (3):
  - Krankenanstalt Rudolfstiftung /ID# 166804, Vienna, Vienna
  - LKH-Univ. Klinikum Graz /ID# 166802, Graz
  - Klinikum Wels - Grieskirchen /ID# 158017, Wels
- Belgium (23):
  - UZ Brussel /ID# 154218, Jette, Brussels Capital
  - Cliniques Universitaires Saint Luc /ID# 154217, Woluwe-Saint-Lambert, Brussels Capital
  - CHU de Liege /ID# 154220, Liège, Liege
  - UZ Gent /ID# 154221, Ghent, Oost-Vlaanderen
  - CLIDERM Bruxelles /ID# 154232, Anderlecht
  - PP Anderlecht /ID# 154230, Anderlecht
  - CHIREC- City Clinic Louise /ID# 154227, Brussels
  - ULB Erasme /ID# 154216, Brussels
  - UZ Antwerp /ID# 154219, Edegem
  - Boonen, Geel, BE /ID# 154233, Geel
  - Coenen, Hasselt, BE /ID# 154234, Hasselt
  - Polyclinique de Herstal /ID# 154226, Herstal
  - Meuleman, Lede, BE /ID# 154238, Lede
  - Grand Hopital de Charleroi /ID# 154222, Loverval
  - Lanssens MD Maldegem BE /ID# 154237, Maldegem
  - C.H.U.de Mons Borinage /ID# 154215, Mons
  - Dr. Pierre-Dominique Ghislain, Mons, BE /ID# 154228, Mons
  - CHU UCL Namur /ID# 154223, Namur
  - CHU UCL Namur /ID# 154224, Namur
  - Ctr Hosp du Bois de l'Abbaye /ID# 154235, Seraing
  - Lecuyer, Thuin, Belgium /ID# 154229, Thuin
  - AZ Sint-Rembert Ziekenhuis /ID# 154231, Torhout
  - Centre Medical 4 sapins /ID# 154236, Wavre
- Czechia (3):
  - Sanatorium, s.r.o /ID# 163593, Chotoviny
  - Vojenska nemocnice /ID# 163592, Olomouc
  - Kozni sanatorium /ID# 163591, Prague
- Kurzen, Freising, DE /ID# 153913, Freising, Germany
- Greece (10):
  - University General Hospital Attikon /ID# 156761, Athens, Attica
  - General Uni hosp of Larissa /ID# 156734, Larissa, Thessaly
  - Duplicate_General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens P /ID# 156762, Athens
  - 251 Airforce General Hospital /ID# 156731, Athens
  - Genl Hospital Andreas Syggros /ID# 156759, Athens
  - Genl Hospital Andreas Syggros /ID# 156760, Athens
  - University Gen Hosp of Patra /ID# 156735, Pátrai
  - General Hospital of Thessaloni /ID# 156728, Thessaloniki
  - General Hospital of Thessaloniki George Papanikolaou /ID# 156758, Thessaloniki
  - 401 GSNA - 401 Army Gen Hosp /ID# 156729, Αthens
- Hungary (8):
  - Miskolci Semmelweis Korhaz es /ID# 153175, Miskolc, Borsod-Abauj Zemplen county
  - Pecsi Tudomanyegyetem /ID# 152612, Pécs, Pecs
  - Markusovszky Egyetemi Oktatókórház /ID# 152616, Szombathely, Vas County
  - Semmelweis Egyetem /ID# 152613, Budapest
  - Debreceni Egyetem Klinikai Központ /ID# 152615, Debrecen
  - Somogy Megyei Kaposi Mor Oktat /ID# 160782, Kaposvár
  - Bacs-Kiskun Megyei Korhaz /ID# 153180, Kecskemét
  - Szegedi Tudomanyegyetem /ID# 152614, Szeged
- Ireland (5):
  - South Infirmary Victoria Univ /ID# 151095, Cork
  - St Vincent's University Hosp /ID# 151084, Dublin
  - Adelaide and Meath Hosp,IE /ID# 151096, Dublin
  - Galway University Hospital /ID# 151097, Galway
  - University Hospital Waterford /ID# 153191, Waterford
- Israel (6):
  - Rabin Medical Center /ID# 149530, Petakh Tikva, Tel Aviv
  - Tel Aviv Sourasky Medical Ctr /ID# 149528, Tel Aviv, Tel Aviv
  - HaEmek Medical Center /ID# 164387, Afula
  - Rambam Health Care Campus /ID# 149529, Haifa
  - Hadassah University Hospital /ID# 149532, Jerusalem
  - Sheba Medical Center /ID# 149531, Ramat Gan
- Lebanon (5):
  - Rizk Hospital /ID# 166027, Beirut
  - Saint Georges Hosp Med Cent /ID# 166024, Beirut
  - American Uni of Beirut Med Cen /ID# 166026, Beirut
  - Trad Hospital and Medical Cent /ID# 166025, Beirut
  - C/O Hotel Dieu de France /ID# 166028, Beirut
- Slovenia (4):
  - General Hospital Celje /ID# 164673, Celje
  - Univ Medical Ctr Ljubljana /ID# 164671, Ljubljana
  - University Medical Ctr Maribor /ID# 164672, Maribor
  - GH Novo Mesto /ID# 164674, Novo Mesto
- Switzerland (3):
  - Hopitaux Universitaires de Geneve /ID# 160090, Geneva, Canton of Geneva
  - Inselspital, Universitaetsklinik /ID# 160089, Bern
  - University Hospital Zurich /ID# 160091, Zurich
- Marmara University Med Faculty /ID# 157903, Istanbul, Turkey (Türkiye)
- United Kingdom (11):
  - Whipps Cross Univ Hospital /ID# 150195, London, London, City of
  - NHS Lanakshire (Monklands) /ID# 152885, Airdire
  - Belfast City Hospital /ID# 168411, Belfast
  - Univ Hospitals Birmingham NHS Foundation trust /ID# 152884, Birmingham
  - Heartlands Hospital /ID# 168409, Birmingham
  - Ninewells Hospital /ID# 168410, Dundee
  - Hull and East Yorkshire NHS /ID# 168413, Hull
  - St. James University Hospital /ID# 150200, Leeds
  - St. John's Institute of Dermat /ID# 150197, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust' /ID# 150199, Newcastle upon Tyne
  - Norfolk and Norwich Univ Hosp /ID# 168412, Norwich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-769.pdf